CLINICAL TRIAL: NCT00760773
Title: Impact of Emergency Department Probiotic Treatment of Diarrheal Illness on Daycare Attendance: Randomized Controlled Trial and Economic Analysis
Brief Title: Impact of Emergency Department Probiotic Treatment of Diarrheal Illness on Daycare Attendance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended and fewer than required number of patients enrolled.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stephen Freedman, Adjunct Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000012686
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis
Keywords: Probiotic treatment; Daycare attendance; Pediatric; Emergency department
MeSH Terms: conditions — Gastroenteritis; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Lacidophil (experimental high dose)
- 2 (Experimental)
  Interventions: Drug: Lacidophil (experimental standard dose)
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lacidophil (experimental high dose) — Each sachet will contain a minimum of 4 billion CFU/sachet. The total weight of all ingredients is 1 gm. All patients in this arm of the study will take 1 sachet twice daily for 5 days. Doses should be ideally separated by 12 hours (minimum of 8 hours) and taken within 30 minutes of food/drink. If the child vomits within 15 minutes of medication administration (initial or subsequent dose), the dose will be repeated. Subjects in this arm will receive the high dose which will consist of 4 billion CFU (1 active sachet) PO BID (total daily dose = 8 billion CFU) x 5 days.
  Arms: 1
Drug: Lacidophil (experimental standard dose) — Each sachet will contain a minimum of 4 billion CFU/sachet. The total weight of all ingredients is 1 gm. All patients in this arm of the study will take 1 sachet twice daily for 5 days. Doses should be ideally separated by 12 hours (minimum of 8 hours) and taken within 30 minutes of food/drink. If the child vomits within 15 minutes of medication administration (initial or subsequent dose), the dose will be repeated. Subjects in this arm will receive the standard dose which will consist of 4 billion CFU (1 active sachet) PO QAM (total daily dose = 4 billion CFU) plus 1 placebo sachet PO QHS x 5 days.
  Arms: 2
Drug: Placebo — The total weight of all ingredients is 1 gm. All patients in this arm of the study will take 1 sachet twice daily for 5 days. Doses should be ideally separated by 12 hours (minimum of 8 hours) and taken within 30 minutes of food/drink. If the child vomits within 15 minutes of medication administration (initial or subsequent dose), the dose will be repeated.
  Arms: 3

SUMMARY:
The objective of this study is to determine for previously healthy children, who present to an ED with acute gastroenteritis, if the probability of daycare absenteeism is significantly different in those who receive a probiotic agent compared to those who receive placebo.

DETAILED DESCRIPTION:
Gastroenteritis in children utilizes significant health care resources and has a significant impact on children, caregivers and society. In the United States, gastroenteritis accounts for more than 1.5 million outpatient visits and 200,000 hospitalizations per year. Data from British Columbia indicate that gastroenteritis annually accounts for 12 million missed workdays by adults and 10 million missed school days by children in this province alone. Canadian data, including the cost of work absenteeism, report the mean annual cost/gastroenteritis case to be $1,089.

Although medications have not routinely been recommended, acute gastroenteritis in children can result in significant morbidity. Thus, physicians and caregivers desire treatment options to reduce the burden of disease. Recently, ondansetron, an antiemetic agent has been found to be effective in pediatric gastroenteritis, and is now frequently employed to reduce vomiting. Probiotics agents may represent another valuable treatment option. Since the early 1990s, research has been conducted on the effects of probiotics, defined as viable microbial preparations that have a beneficial effect on the health and well being of the host.

A recent Cochrane Database systematic review recently concluded that "probiotics appear to be a useful adjunct to rehydration therapy in treating acute, infectious diarrhea." However, the review also concluded that more research is needed to determine which specific probiotic regimens should be employed in specific patient groups. The later statement is of particular importance in North America as probiotics are not a mainstay of clinical practice. While only 18% of Canadian physicians are aware of research on probiotics, 82% feel that more probiotic research is needed, and 76% feel there is a role for probiotics in their practice. This discrepancy likely is due to the absence of probiotic trials in North American patients and because the outcome measures evaluated often have had limited clinical applicability. Since most episodes of acute diarrhea require no specific treatment, cost-effectiveness analyses are also required before the widespread use of probiotics can be endorsed.

ELIGIBILITY:
Inclusion Criteria:

* Acute gastroenteritis as determined by the supervising physician.
* Attend daycare
* Presence of diarrhea.
* Duration of vomiting or diarrhea less than 96 hours.
* Age greater than 90 days
* Age less than 48 months

Exclusion Criteria:

* Presence of an indwelling vascular access line or congenital heart disease.
* Taking immunosuppressive therapy or history of immunodeficiency (including all primary, secondary and acquired states)
* Have recently had cardiac, oral or gastrointestinal surgery
* Pancreatic dysfunction or bloody diarrhea
* History of: hematochezia, underlying chronic gastrointestinal problem, short bowel syndrome or inflammatory bowel disease
* Family member with an indwelling vascular access line, on immunosuppressive therapy or with a known immunodeficiency
* Undergoing radiation therapy
* Exclusively breastfed
* Bilious or bloody vomitus
* Previously enrolled in this trial
* Inability to speak or read English

Ages: 4 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2009-04; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children missing a day of daycare related to vomiting, diarrhea, dehydration, fever, or fluid refusal. | 2 weeks

SECONDARY OUTCOMES:
Return visits for unscheduled care to a health care provider related to vomiting, diarrhea, dehydration, fever, or fluid refusal. | 2 weeks
Intravenous rehydration | 2 weeks
Duration of diarrhea | Meaured by outcome
Duration of vomiting | Meaured by outcome
Number of days the child does not go to daycare. | Measured by outcome
Work absenteeism | 2 weeks
Economic analysis | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte Justine, Montreal, Quebec